CLINICAL TRIAL: NCT01412359
Title: Compassionate Use of Omegaven® in the Treatment of Parenteral Nutrition Associated Hepatic Injury
Status: Approved for marketing | Type: Expanded Access
Sponsor: Jeffrey Rudolph (Other)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Sponsor-Investigator, Jeffrey Rudolph, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Other Study IDs: PRO08080394
Record Dates: First submitted 2011-08-02; First posted 2011-08-09 (Estimated); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Total Parenteral Nutrition-induced Cholestasis
Keywords: TPN Cholestasis
MeSH Terms: interventions — fish oil triglycerides

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Omegaven® — Omegaven® 10% fat emulsion 1g/kg/day to infuse via IV over a period of 12 -24 hours every day until patient no longer requires intravenous lipid emulsion, is determined ineffective, or the patient stops participating in the study for any reason.
  Other Names: Intavenous fish oil emulsion

SUMMARY:
The overall purpose of this study is to determine if replacing standard soybean oil based fat emulsions with Omegaven®, a fish oil based fat emulsion, can reverse or prevent the progression of parenteral nutrition associated cholestasis. It is a compassionate use protocol for patients who already have significant cholestasis related to parenteral nutrition.

DETAILED DESCRIPTION:
In the United States, patients dependent upon parenteral nutrition (PN) receive parenteral fat emulsions composed of soybean oils. Lipids are necessary in PN dependent patients due to their high caloric value and essential fatty acid content. Phytosterols such as those contained in soybean oil based fat emulsions are thought to have a deleterious effect on biliary secretion and they have been implicated in predisposing patients to PN associated liver disease. Children requiring prolonged courses of PN are at risk for developing PN associated liver disease. The investigators hypothesize that although soybean oil based fat emulsions prevent fatty acid deficiency, they are not cleared in a manner similar to enteral chylomicrons and therefore accumulate in the liver resulting in steatotic liver injury.

Animal studies have shown that fish oil based IV fat emulsions(IFE)which are high in eicosapentaenic and docosahexaenoic acid, reduce impairment of bile flow seen in cholestasis caused by conventional fat emulsions. Omegaven® is a fish oil based IV fat emulsion. The investigators hypothesize that administering Omegaven® in place of conventional soybean fat emulsions may reverse or prevent the progression of PN associated cholestasis and thus allow the patient to be maintained on adequate PN until he/she is able to ingest adequate nutrition enterally.

Primary outcome measures to be addressed include the normalization of liver enzymes including bilirubin upon the start of Omegaven® and continued growth on Omegaven®. Safety measures will include the prevalence of essential fatty acid deficiency, hypertriglyceridemia, and bleeding disorders.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 2 months -10 years of age.
* Patients who are PN dependent (unable to meet nutritional needs solely by enteral nutrition) and are expected to require PN for at least another 30 days
* Patients considered eligible for study participation must have parenteral nutrition associated liver disease (PNALD) as defined by a direct bilirubin of >2.0mg/dL. Other causes of liver disease should be excluded. A liver biopsy is not necessary for treatment.
* 2 consecutive direct bilirubin test results >2.0mg/dL
* The patient must have failed standard therapies to prevent the progression of liver disease such as surgical treatment, cyclic TPN, avoiding overfeeding, reduction/removal of copper and manganese from TPN, advancement of enteral feeding, and use of ursodiol (Actigall).
* Subjects who are currently under treatment for PNALD with Compassionate Use Omegaven and have a direct Bilirubin of< 2, but who remain TPN dependent and require continued therapy with Omegaven.

Exclusion Criteria:

* Other known causes of chronic liver disease (hepatitis C, cystic fibrosis, biliary atresia and alpha 1 anti-trypsin deficiency)
* Enrollment in any other clinical trial involving an investigational agent (unless approved by the designated physicians on the multidisciplinary team)
* The parent, guardian, or child is unwilling to provide consent or assent
* Allergy to any fish product, egg protein, and/or previous allergy to Omegaven
* Active coagulopathies characterized by on-going bleeding or by a requirement for clotting factor replacement such as fresh frozen plasma or cryoprecipitate to maintain homeostasis
* Impaired lipid metabolism or severe hyperlipidemia with or without pancreatitis
* Unstable diabetes mellitus
* Stroke/embolism
* Collapse and shock
* Undefined coma status
* Active infection at time of initiation of Omegaven® up until such time as child is afebrile with stable vital signs and one negative 48 hour culture.

Ages: 2 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A Rudolph, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania, United States